CLINICAL TRIAL: NCT04077476
Title: Feasibility of Online Yoga Plus Social Support to Improve Elevated PTS in Mothers Who Have Experienced Stillbirth
Brief Title: Feasibility of Online Yoga With Facebook After Stillbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00010215
Record Dates: First submitted 2019-06-18; First posted 2019-09-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Stillbirth; Post-traumatic Stress Disorder; Anxiety; Depression
MeSH Terms: conditions — Stillbirth; Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: The study design is a randomized control trial with baseline and post-intervention (8 wks from baseline) assessments. Participants are randomized into either an online yoga group or an online yoga plus Facebook group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Yoga (Active Comparator): Participants in both groups will follow a prescription of classes the research team (including a 200-hour yoga instructor) developed, and is safe and appropriate for this study population. The yoga prescription will be based on the prescription used in the current R34 study (see reference for description), and modified based on results (i.e., participant feedback). Participants will be given instructions about how to use the online yoga class platform (Udaya) during the intake appointment.
  Interventions: Behavioral: Online Yoga
- Online Yoga + Facebook (Experimental): In addition to what is described above, participants will be provided instructions on how to join the private Facebook group. The Facebook group will be an informal platform where participants can connect with other people in the online + SN group to share their experiences with yoga as it relates to their stillbirths. Current social media intervention research suggests careful consideration must be given to the intervention. The current intervention will be designed based on results of focus groups asking stillbirth moms who have completed an online yoga intervention what they would find helpful in a Facebook intervention. For instance, preferences included having a moderator, rules about what they can post (e.g., no "rainbow babies"), and discussion about both stillbirth and life in general.
  Interventions: Behavioral: Online Yoga + Facebook

INTERVENTIONS:
Behavioral: Online Yoga + Facebook — Each week, the research team will post a prompt for discussion to encourage participation. Prompts will be developed in the beginning stages of the project based on data from the current R34 study and with guidance from consultant Waibel. Participants will be encouraged to post about their experiences with the intervention and stillbirth (emotional support), share resources, (informational support), and offer feedback and advice (appraisal support). Participants will not be required to adhere to certain criteria for engagement (e.g., number of posts, etc.), other than their weekly log in. This is to account for different types of engagement when using social networking as a means of support (e.g., posting, just reading); the benefits of each type of engagement are person-specific. The page will be moderated by members of the research team, who will post prompts and ensure content is updated and appropriate. No members can be added to the group without approval from the research team.
  Arms: Online Yoga + Facebook
Behavioral: Online Yoga — Participants will complete a series of videos covering basic poses and safety techniques, tracked using the Wistia plugin software. Once complete, they will be able to access the library of pre-selected classes (range in time from 10-90 minutes). Participants will be asked to complete at least 60 minutes of yoga per week; participants may choose any classes to yield 60 minutes. Preliminary data from the current R34 study suggests 60 minutes is a feasible amount of time for yoga participation. There is no upper limit to the number of minutes participants can complete.
  Arms: Online Yoga

SUMMARY:
The purpose of this study is to investigate the feasibility and effectiveness on PTSD symptoms of the addition of a Facebook group to an online yoga intervention for women following a stillbirth.

DETAILED DESCRIPTION:
Each year in the United States, over 26,000 women experience a stillbirth (death of a fetus ≥20 weeks of gestation). Stillbirth moms are six times more likely to develop post-traumatic stress disorder (PTSD) and four times more likely to have anxiety and depressive symptoms than moms who have live births. Stillbirth moms also experience poor sleep, lack of support, and disenfranchised grief. The negative effects of a stillbirth may last for years and may negatively impact subsequent pregnancies; many get pregnant within a year after their loss.

There is currently no standard of care for women who have experienced a stillbirth. Recommended treatment after a stillbirth typically includes medication and referral to support groups and therapists. While medication may be helpful to some women, others may be averse to medication. Support groups, if not catered to bereaved moms, may trigger post-traumatic stress symptoms. Other barriers may inhibit participation in outside the home treatment after stillbirth, such as seeing babies or having to explain their stillbirths, as reported in one study.

Yoga may be a complementary strategy to help mothers cope with post-traumatic stress. Evidence suggests yoga may improve physical and mental health (e.g., anxiety, depressive symptoms) in various populations who experience trauma (e.g., war veterans, abuse victims). Research suggests those who participate in yoga are likely to exhibit healthier behaviors (i.e., physical activity, healthy diet, abstain from alcohol/substance abuse). Yoga is safe and feasible for pregnant and post-partum women. Although yoga may be an effective strategy for PTSD following a stillbirth, due to the barriers these mothers experience, attending yoga classes at a studio may not be feasible.

Online interventions are growing in popularity and may be a way to overcome barriers to participation in treatment for stillbirth moms. Investigators are currently conducting a feasibility study to explore the use of online yoga to improve PTSD in stillbirth moms (NIH#R34AT008808). Data collection will be complete in May, 2019. Supplemental to this study, investigators conducted interviews with stillbirth moms who have finished the intervention. A brief view of the data from these interviews suggest women liked the online platform but felt isolated and wanted more social interaction during the intervention.

When an intervention is delivered online (e.g., through social networking: engaging in social interactions though online platforms), the natural social interaction that happens during in-person interventions is lacking. Research suggests giving and receiving support is an adaptive coping strategy to reduce PTSD symptoms, anxiety, and depressive symptoms. Stillbirth moms who perceived adequate levels of social support had significantly lower anxiety and depression levels than those who did not. There is a need to explore the feasibility of online interventions that include social networking to determine the relationship between online interventions and social support, and how social support acts as a mediator between social networking and PTSD, anxiety, depressive symptoms, and health behaviors.

Interventions that include a Facebook component have been shown to effectively improve social support, however little is known about the optimal structure of this type of intervention. One research study asserts existing social media platforms (e.g., Facebook) as ideal because members are familiar with the platform's social norms (e.g., how to post, "like," and comment). There is a need to explore the feasibility of a social networking component (i.e., Facebook) in addition to an online yoga intervention and the effects this might have on social support as well as PTSD, anxiety, depressive symptoms and health behaviors.

Therefore, the purpose of this study is to:

1. Examine the feasibility (acceptability, demand) of a social networking component (i.e., Facebook) to an eight-week online yoga intervention for a future U01 application.
2. Explore the preliminary effects (i.e., not powered for effects) of a social networking component (i.e., Facebook) added to an eight-week online yoga intervention on social support.
3. Explore the mechanism (i.e., social support) by which social networking may impact PTSD symptoms, anxiety, depressive symptoms and health behaviors (i.e., physical activity, diet, smoking, and alcohol consumption).

ELIGIBILITY:
Inclusion Criteria:

* Women
* Ages 18+
* Had a stillbirth within the past 3 years
* Can safely participate in exercise as determined by the Physical Activity Readiness Questionnaire (PAR-Q): Answer "no" to all items on PAR-Q (can participate safely)
* Not currently practicing yoga: Operationally defined as participating ≥60 minutes per week within the past 6 months
* Have symptoms of PTSD (>24 on the Impact of Events Scale-Revised (IES-R), which is classified as "PTSD is a clinical concern."
* Not pregnant at the time of the intervention
* Have, or be willing to create, a Facebook account
* Willing to be randomized
* Able to read and understand English

Exclusion Criteria:

* Unstable psychiatric condition (score of 20-27 on the Patient Health Questionnaire (PHQ-9)), determined by a licensed clinical social worker
* Suicidal ideation (answer 1, 2, or 3 on the last question of the PHQ-9), determined by a licensed clinical social worker
* Previous participation in a study by the research team

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Berlin Social Support Scale | Change from baseline (week 0) to post (week 8)
  The Berlin Social Support Scale is a 17-item inventory used to assess social support. The scale consists of 4 subscales: emotional support, instrumental support, need for support, and support seeking. The questions are rated on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree).
Feasibility: satisfaction survey | Post (week 8)
  Researcher-developed surveys are used to assess feasibility with questions related to satisfaction, acceptability, and demand of both study arms. Items are rated on a 5-point Likert scale ranging from 1 (lowest) to 5 (highest).
Impact of Events Scale-Revised | Change from baseline (week 0) to post (week 8)
  The Impact of Events Scale-Revised (IES-R) is a 22-item inventory used to assess symptoms of post-traumatic stress disorder. The scale contains items pertaining to a person's (direct or indirect) response to a traumatic event within the past week (e.g., "I had trouble staying asleep."). The items are rated on a 5-point Likert scale from 0 (never) to 4 (extremely).
State-Trait Anxiety Inventory | Change from baseline (week 0) to post (week 8)
  The State-Trait Anxiety Inventory is a 40-item inventory used to assess symptoms of anxiety. The two subsections of the inventory are state-specific and trait-specific. Each item is rated on a 4-point scale from 1 (not at all) to 4 (very much so).
Patient Health Questionnaire (PHQ-9) | Change from baseline (week 0) to post (week 8)
  The Patient Health Questionnaire (PHQ-9) is a 9-item inventory used to assess depressive symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day).

SECONDARY OUTCOMES:
National Cancer Institute's Multifactor Screener (diet) | Change from baseline (week 0) to post (week 8)
  The National Cancer Institute's Multifactor Screener is a 16-item inventory used to assessed diet. It contains questions about how often respondents eat and drink certain foods or drinks. Items are rated on a 9-point Likert scale with "Never" and "4 or more times per day" as anchors.
International Physical Activity Questionnaire | Change from baseline (week 0) to post (week 8)
  The International Physical Activity Questionnaire (IPAQ) is a 7-item inventory used to assess physical activity. Each item asks about time spent doing certain activities within the past week. Responses can range from 0 (not at all) to 7 days per week and/or 24 hours per day. Responses are recorded in days per week and hours/minutes per day. Higher numbers of days per week and/or hours/minutes per day indicate higher levels of physical activity.
Smoking/Alcohol Behavior | Change from baseline (week 0) to post (week 8)
  One-item questions regarding smoking alcohol consumption are used to assess smoking behavior and alcohol consumption. The items ask how many drinks per day/week participants consume and how much they smoke per day/week, if at all. Higher numbers indicate a higher frequency of each behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona Biomedical Collaborative, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Blackmore ER, Cote-Arsenault D, Tang W, Glover V, Evans J, Golding J, O'Connor TG. Previous prenatal loss as a predictor of perinatal depression and anxiety. Br J Psychiatry. 2011 May;198(5):373-8. doi: 10.1192/bjp.bp.110.083105. Epub 2011 Mar 3. PMID 21372060
- [Result] Hughes PM, Turton P, Evans CD. Stillbirth as risk factor for depression and anxiety in the subsequent pregnancy: cohort study. BMJ. 1999 Jun 26;318(7200):1721-4. doi: 10.1136/bmj.318.7200.1721. PMID 10381705
- [Result] Ellis A, Chebsey C, Storey C, Bradley S, Jackson S, Flenady V, Heazell A, Siassakos D. Systematic review to understand and improve care after stillbirth: a review of parents' and healthcare professionals' experiences. BMC Pregnancy Childbirth. 2016 Jan 25;16:16. doi: 10.1186/s12884-016-0806-2. PMID 26810220
- [Result] Mitchell KS, Dick AM, DiMartino DM, Smith BN, Niles B, Koenen KC, Street A. A pilot study of a randomized controlled trial of yoga as an intervention for PTSD symptoms in women. J Trauma Stress. 2014 Apr;27(2):121-8. doi: 10.1002/jts.21903. Epub 2014 Mar 25. PMID 24668767
- [Result] Park CL, Riley KE, Bedesin E, Stewart VM. Why practice yoga? Practitioners' motivations for adopting and maintaining yoga practice. J Health Psychol. 2016 Jun;21(6):887-96. doi: 10.1177/1359105314541314. Epub 2014 Jul 16. PMID 25030795
- [Result] Buttner MM, Brock RL, O'Hara MW, Stuart S. Efficacy of yoga for depressed postpartum women: A randomized controlled trial. Complement Ther Clin Pract. 2015 May;21(2):94-100. doi: 10.1016/j.ctcp.2015.03.003. Epub 2015 Apr 1. PMID 25886805
- [Result] Naslund JA, Aschbrenner KA, Marsch LA, Bartels SJ. The future of mental health care: peer-to-peer support and social media. Epidemiol Psychiatr Sci. 2016 Apr;25(2):113-22. doi: 10.1017/S2045796015001067. Epub 2016 Jan 8. PMID 26744309
- [Result] McAlpine H, Joubert L, Martin-Sanchez F, Merolli M, Drummond KJ. A systematic review of types and efficacy of online interventions for cancer patients. Patient Educ Couns. 2015 Mar;98(3):283-95. doi: 10.1016/j.pec.2014.11.002. Epub 2014 Nov 18. PMID 25535016
- [Result] Cacciatore J, Schnebly S, Froen JF. The effects of social support on maternal anxiety and depression after stillbirth. Health Soc Care Community. 2009 Mar;17(2):167-76. doi: 10.1111/j.1365-2524.2008.00814.x. PMID 19281517
- [Result] Cavallo DN, Tate DF, Ries AV, Brown JD, DeVellis RF, Ammerman AS. A social media-based physical activity intervention: a randomized controlled trial. Am J Prev Med. 2012 Nov;43(5):527-32. doi: 10.1016/j.amepre.2012.07.019. PMID 23079176
- [Derived] Sullivan M, Huberty J, Green J, Cacciatore J. Adding a Facebook Support Group to an Online Yoga Randomized Trial for Women Who Have Experienced Stillbirth: A Feasibility Study. J Integr Complement Med. 2022 Feb;28(2):179-187. doi: 10.1089/jicm.2021.0097. Epub 2022 Jan 11. PMID 35167361